CLINICAL TRIAL: NCT03792269
Title: An Open-label, Randomized, Phase II Clinical Trial Comparing the Efficacy and Safety of Intraperitoneal and System Chemotherapy Versus XELOX as First-line Chemotherapy for Metastatic Colorectal Cancer
Brief Title: Intraperitoneal and System Chemotherapy Versus XELOX as First-line Chemotherapy for mCRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jing Hu, investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mCRC-PC
Record Dates: First submitted 2019-01-01; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Cancer Metastatic; Chemotherapy Effect; Chemotherapeutic Toxicity
MeSH Terms: interventions — Irinotecan; Oxaliplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-channel chemotherapy (Experimental): Patients will receive intraperitoneal irinotecan (50mg, d1, q2w).
  Interventions: Drug: Irinotecan
- Control Group (Active Comparator): Patients will receive intravenous oxaliplatin (130mg/m^2, d1, q3w), and oral capecitabine (1.0g, d1-14, q3w).
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Irinotecan — intraperitoneal
  Arms: Multi-channel chemotherapy
Drug: Oxaliplatin — intravenous
  Arms: Control Group
Drug: Capecitabine
  Other Names: Oral
  Arms: Control Group

SUMMARY:
XELOX as first-line treatment regimen has limited efficacy against patients with metastatic colorectal cancer (mCRC). Peritoneal metastasis is one of the most lethal factor for mCRC. Intraperitoneal chemotherapy has became a widely accepted strategy in the treatment of peritoneal dissemination. We hypothesized that combined multi-channel administration, such as intraperitoneal chemotherapy, oral chemotherapy, and intravenous chemotherapy, can produce better results than XELOX for first-line treatment for mCRC patients.

ELIGIBILITY:
Inclusion Criteria:

Patients must have histologically confirmed adenocarcinoma of clorectal with inoperable locally advanced or metastatic disease, not amenable to curative therapy.

Patients must have measurable disease, according to the Response Evaluation Criteria in Solid Tumors (RECIST, v1.1), assessed using imaging techniques (CT or MRI).

Women of childbearing potential must be non-pregnant (negative pregnancy test within 72 hours prior to chemotherapy, postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential) and nonlactating, and men and women must be willing to exercise an effective form of birth control (abstinence/contraception) while on study and for 6 months after therapy completed Eastern Cooperative Oncology Group (ECOG) Performance status 0, 1 or 2. Absolute neutrophil count (ANC) >=1,500/ul Platelets (PLT) >=75,000/ul Serum bilirubin <= 1.5 × upper limit of normal (ULN) Aspartate transaminase (AST) or alanine aminotransferase (ALT) <= 2.5 × ULN (or <= 5 × ULN in patients with liver metastases) Alkaline phosphatase <= 2.5 × ULN (or <= 5 × ULN in patients with liver metastases, or <= 10 × ULN in patients with bone but no liver metastases) Albumin >= 25 g/L. Creatinine clearance >= 60 mL/min. Life expectancy of at least 3 months. Signed informed consent.

Exclusion Criteria:

Previous chemotherapy for advanced/metastatic disease (prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrolment into the study).

Patients with active (significant or uncontrolled) gastrointestinal bleeding. Residual relevant toxicity resulting from previous therapy (with the exception of alopecia), e.g. neurological toxicity ≥ grade 2 NCI-CTCAE 4.0.

Other malignancy within the last 5 years, except for carcinoma in situ of the cervix, or basal cell carcinoma.

History of documented congestive heart failure; angina pectoris requiring medication;evidence of transmural myocardial infarction on ECG; poorly controlled hypertension (systolic BP > 180 mmHg or diastolic BP > 100 mmHg); clinically significant valvular heart disease; or high risk uncontrollable arrhythmias.

Baseline left ventricular ejection fraction (LVEF) < 50% (measured by echocardiography or MUGA).

Patients with dyspnoea at rest due to complications of advanced malignancy or other disease, or who require supportive oxygen therapy.

Patients receiving chronic or high dose corticosteroid therapy. (Inhaled steroids and short courses of oral steroids for anti-emesis or as an appetite stimulant are allowed).

Clinically significant hearing abnormality. Known dihydropyrimidine dehydrogenase (DPD) deficiency. History or clinical evidence of brain metastases. Serious uncontrolled systemic intercurrent illness, e.g. infections or poorly controlled diabetes.

Positive serum pregnancy test in women of childbearing potential. Received any investigational drug treatment within 4 weeks of start of study treatment.

Radiotherapy within 4 weeks of start of study treatment (2 week interval allowed if palliative radiotherapy given to bone metastatic site peripherally and patient recovered from any acute toxicity;prior adjuvant radiotherapy is allowed if complete at least 6 months ).

Major surgery within 4 weeks of start of study treatment, without complete recovery.

Patients with known active infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV).

Known hypersensitivity to any of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to 1 year
  PFS is the period between the first course of treatment to disease recurrence. The follow-up work will be performed every 6 weeks until disease recurrence or loss to follow-up.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 2 years
  OS is the period between the first course of treatment to death. The follow-up work will be performed every 3 months until death or loss to follow-up.
Objective Response Rate (ORR) | up to 24 weeks
  CT/MRI will be performed every 2 cycles of treatment for short-term efficacy. evaluation
Adverse Events (AE) | up to 2 years
  Adverse effects will be recorded during the whole treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jing, Study Chair — The Comprehensive Cancer Center of Nanjing Drum Tower Hospital
Locations (1):
- The Comprehensive Cancer Center of Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No